CLINICAL TRIAL: NCT05453435
Title: Entecavir Prophylaxis for Hepatitis B Reactivation for CD20 Positive B-cell Lymphoma Patients With Resolved Hepatitis B (Negative Hepatitis B Surface Antigen, Positive Hepatitis B Core Antibody) (REHEB)：a Single Arm, Open Label, Multi-center Phase II Study
Brief Title: Entecavir Prophylaxis for Hepatitis B Reactivation for CD20 Positive B-cell Lymphoma Patients With Resolved Hepatitis B (Negative Hepatitis B Surface Antigen, Positive Hepatitis B Core Antibody)
Acronym: REHEB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-352-01
Record Dates: First submitted 2022-07-02; First posted 2022-07-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Resolved Hepatitis B; CD20 Positive B-cell Lymphoma
MeSH Terms: interventions — entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Entecavir prophylaxis (Experimental): 0.5mg qd
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — All patients enrolled in the study will accept entecavir prophylaxis that initiates within 1 week before the first course of CD20 monoclonal antibody therapy, and continues until 6 months after completing CD20 monoclonal antibody therapy.

SUMMARY:
This phase 2 trial aims to evaluate the efficacy of entecavir prophylacxis for hepatitis B virus (HBV) reactivation that continues until 6 months after completing CD20 monoclonal antibody therapy in patients with CD20-positive B-cell lymphomas and resolved hepatitis B (negative hepatitis B surface antigen, positive hepatitis B core antibody).

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed CD20 positive B-cell lymphoma;
* Plan to receive first-line anti-lymphoma therapy containing CD20 monoclonal antibodies;
* Negative HBsAg, HBV-DNA lower than the detection limit and positive anti-HBC at baseline;
* Total bilirubin less than 1.5X the upper limit of normal (ULN), AST and ALT less than 2.5X ULN;
* ECOG PS: 0~2;
* Estimated survival time >3 months.

Exclusion Criteria:

* Positive HBsAg or HBV-DNA higher than the detection limit at baseline;
* Previous chemotherapy or radiotherapy for lymphoma;
* Other primary liver diseases, such as chronic hepatitis C, hepatitis D, autoimmune hepatitis, Wilson' s disease or primary biliary cirrhosis;
* Pregnant or lactating women;
* History of immunodeficiency, including positive HIV, or other acquired congenital immunodeficiency disease, or history of organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cumulative HBV reactivation rate | 12 months
  Cumulative incidence of hepatitis B virus reactivation

SECONDARY OUTCOMES:
Incidence of HBV-related liver failure | 12 months
  Incidence of HBV-related liver failure
Incidence of HBV-related chemotherapy disruption | 12 months
  Incidence of HBV-related chemotherapy disruption

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, State..., China